CLINICAL TRIAL: NCT01877603
Title: The Relation Between Plasma Irisin Level and Endothelial Dysfunction in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Other Study IDs: 2013Wze030
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Irisin; Endothelial Dysfunction; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- type 2 diabetes: We select 200 newly diagnosed type 2 diabetic patients. Plasma irisin levels will be measured, and endothelial function will be determined.

SUMMARY:
Irisin is a signaling protein that is released into the blood from skeletal muscle after proteolysis of the membrane protein FNDC5 . FNDC5, encoded by the Fndc5 gene. Irisin activity on subcutaneous white adipose tissue, both in culture and in vivo, stimulated UCP1 expression and induction of brown adipocytes in white adipose tissue depots, a process known as white fat ''browning''. Irisin increases total energy expenditure in animal models, and irisin expression in mice fed a high fat diet resulted in a significant improvement in glucose tolerance and a reduction in fasting insulin levels. Collectively, these data suggest that decreased serum irisin levels may be associated with the development of insulin resistance and Type 2 diabetes. Indeed, some studies showed that irisin levels were decreased in newly diagnosed Type 2 diabetes.

Endothelial dysfunction is an early physiological event in atherosclerosis. However, to date, no data are available on the relationship between circulating irisin and endothelial dysfunction in diabetes. Therefore, the investigators hypothesized that circulating irisin level is associated with endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetic patients
* aged 40～70 years

Exclusion Criteria:

* Patients with hypertension and those with micro- and macroangiopathy, including nephropathy [urinary albumin excretion rate (UAER) > 20 μg/min], retinopathy (at least one microaneurysm or hemorrhage or exudates in either eye), neuropathy (pain in extremities, paresthesias, and absent tendon reﬂexes and/or absent vibration sense), coronary artery disease (myocardial infarction, ischemia electrocardiogram changes, and angina), cerebrovascular disease (transient ischemic attack or stroke), and peripheral vascular disease (the abolition of one or more peripheral arterial pulse and/or intermittent claudication and/or a past history of revascularization of the lower limbs) were excluded from the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From July 2013 to Dec 2013, a total of 200 Chinese Han newly diagnosed type 2 diabetic patients were selected. They had been referred to our hospital and were aged 40～70 years.
  During the same period, 50 healthy subjects (all from medical staff in our hospital) were selected as control subjects.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The relation between plasma irisin and endothelium-dependent vasodilation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China